CLINICAL TRIAL: NCT05539404
Title: French Acute Randomized Controlled Trial Using Multimodal Imaging for Endovascular Treatment of Patients With Large Cerebral Infarction With Substantial Penumbra up to 24 Hours
Brief Title: Evaluate Endovascular Treatment of Large Ischemic Stroke With Substantial Penumbra.
Acronym: FrameLP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study ends for scientific reasons
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/21/0336; 2021-A03139-32 (Other: ID-RCB)
Record Dates: First submitted 2022-07-11; First posted 2022-09-14 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; large stroke; Multimodal brain imaging; Thrombectomy; endovascular treatment
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Strategy Group (Experimental): endovascular treatment in addition to best medical treatment
  Interventions: Procedure: Endovascular treatment in addition of best medical treatment.
- Control Strategy Group (No Intervention): best medical treatment

INTERVENTIONS:
Procedure: Endovascular treatment in addition of best medical treatment. — Endovascular treatment (EVT) of acute ischemic stroke (AIS) related to an anterior large cerebral vessel occlusion (LVO)
  Other Names: Mechanical thrombectomy
  Arms: Experimental Strategy Group

SUMMARY:
Large cerebral infarctions are frequent and associated with a poor outcome. Previous cohort studies results suggest that patients with an acute ischemic stroke with large core and substantial penumbra on perfusion imaging benefit from EVT while those with no salvageable ischemic tissue did not. The Investigator aim to demonstrate in a randomized controlled trials (RCT) that EVT (Endo Vascular Treatment) in addition to BMT (Best Medical Treatment) increases the rate of functional recovery (mRS 0-2) at 3 months in patients with a LVO-related AIS with a large core and substantial penumbra evolving for less than 24hrs

DETAILED DESCRIPTION:
The reperfusion of salvageable ischemic tissue (penumbra) to improve functional recovery is the aim of the endovascular treatment (EVT) of acute ischemic stroke (AIS) complicating large cerebral vessel occlusion (LVO). Downstream of an LVO, imaging profiles are highly variable ranging from a large completed infarction within 2 hrs to a small core and a large mismatch at 24 hrs after onset . A large core is typically associated with a poor prognosis and was a common exclusion criterion from the RCTs that demonstrated the efficacy of EVT for LVO related AIS . However the investigator recently reported that AIS with a large core 1- represent 20% of the LVO-related AIS scanned within 6 hours after onset 2- Up to 50% had a MM on perfusion imaging and 3- EVT increases the rate of functional recovery in patients with a large core over BMT only in the subgroup of patients with a MM (Mismatch) on baseline imaging .

One hundred and eighty patients experiencing an LVO-related AIS within 24 hours after last known well, with a documented large core (>70mL) and a MM on baseline imaging will be randomized (1:1) to undergo EVT+BMT vs. BMT in a multicenter, randomized, controlled, open-label, in parallel groups with blinded endpoint evaluation (PROBE design) superiority trial.

Study participants will be followed up for 6 months. Participants will be treated and managed in acute stroke units by certified stroke neurologists and neurointerventionists according to the current recommendations . Neurological deficit will be assessed using the NIH Stroke Scale (NIHSS) by certified investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing an acute ischemic stroke related to an anterior proximal large vessel occlusion (ICA/M1/Tandem) on MR or CT-angiography evolving for less than 24 hours from last known to be well. For patients experiencing a wake-up stroke or a stroke of unknown onset the mid-point between last seen well and symptoms discovery + the delay between symptoms discovery to randomization, will be used to calculate the delay between symptom onset to randomization.
* On baseline imaging (MRI Diffusion Weighted Imaging/Perfusion Weighted Imaging or CTP) L.P. profile defined by a Large Core > 70 mL, and a MM ratio>1.4 using RAPID software.
* Delay between end of imaging and randomization <90 min.
* Expected delay between end of imaging and femoral puncture < 60 min
* Best medical treatment including IV thrombolysis if indicated
* Surrogate decision maker's consent or emergency inclusion form.
* Affiliated person or beneficiary of a social security scheme.

Exclusion Criteria:

* Pre-Stroke mRS >1.
* Other serious advanced or terminal illness or life expectancy is estimated to be less than 6 months.
* Pre-existing medical, neurological or psychiatric condition that would confound the neurological or functional evaluation.
* Pregnancy and breastfeeding
* Inability to undergo contrast brain perfusion MR or CT.
* Technically inadequate perfusion imaging precluding L.P. profile assessment
* Occlusion in multiple proximal vascular site territories (eg. bilateral anterior circulation occlusion or anterior + posterior circulation occlusions).
* Known allergy to iodine precluding EVT.
* Vessel anatomy or tortuosity precluding EVT.
* Patient under judicial protection.
* Participation in another interventional or therapeutic study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Rate of patients achieving a functional recovery defined by modified Rankin Scale 0-2 at 3 months | 3 months
  Good functional outcome will be defined by a Modified Rankin Scale of 0-2, done by a certified rater, blinded of the arm of the randomization

SECONDARY OUTCOMES:
modified Rankin Scale | 3 and 6 months
  Rate of patients with Modified Rankin Scale of 0-2 , rate of patients with Modified Rankin Scale 0-3 and Global disability assessed by overall distribution of the Modified Rankin Scale (shift analysis combining scores 5 and 6)
National Institute of Health Scale | Day 1
  Rate of patients achieving an early neurological improvement National Institutes of Health Stroke Scale (NIHSS) >or=8 reduction from baseline to day 1 or National Institutes of Health Stroke Scale (NIHSS) =0-1 at day 1
Modified Thrombolysis in Cerebral Infarction score | Day 1
  Rate of successful reperfusion in the EndoVascular Treatment+Best medical treatment arm defined by a mTICI ( Modified Thrombolysis in Cerebral Infarction) 2bc3 score
mortality rate | 3 and 6 months
  Number of subject who die during the study participation in each arm.
Symptomatic Hemorrhagic Transformation | 36 hours
  Symptomatic hemorrhagic transformation is defined by an intra cerebral hemorrhage (European Cooperative Acute Stroke Study III classification " ECASS III ") associated with a 4 or more point increase on the National Institute of Health " NIH " Stroke Scale by comparison with NIH Stroke Scale immediately predeterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc OLIVOT, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (9):
- France (9):
  - Hôpital Pellegrin, Bordeaux
  - University Hospital of Lille Hôpital Roger Salengro, Lille
  - University Hospital of Limoges Hôpital Dupuytren 1, Limoges
  - University Hospital of Montpellier Hôpital Gui de Chauliac, Montpellier
  - University Hospital of Nancy (CHRU) Hôpital central, Nancy
  - Fondation Adolphe de Rothschild Hospital, Paris
  - University Hospital Pitié-Salpétrière AP-HP, Paris
  - Foch Hospital Centre, Suresnes
  - University Hospital Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No